CLINICAL TRIAL: NCT07074366
Title: Personality Traits of TMD Experts Really Matters, A New Era in TMD Management
Brief Title: How Dentists' Personality Traits Affect Communication and Treatment Outcomes in TMD Patients
Acronym: TMD
Status: Completed | Type: Observational
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, Lecturer of Oral and Maxillofacial Surgery, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: RP.25.05.1
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Disorders; Psychological Distress; Chronic Orofacial Pain
Keywords: TMD; Splint Therapy; Dentist Personality; Patient Satisfaction
MeSH Terms: conditions — Temporomandibular Joint Disorders; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMD Patients Assigned to Dentists: Patients diagnosed with TMDs were randomly assigned to dentists with varying personality traits. All patients received standardized splint therapy and were followed for six months. Key patient-reported outcomes-including communication quality, satisfaction with treatment, adherence to splint use, and changes in psychological distress (DASS-10)-were assessed to examine the influence of dentist personality on treatment effectiveness.
  Interventions: Behavioral: Splint Therapy with Structured Communication

INTERVENTIONS:
Behavioral: Splint Therapy with Structured Communication — All participants received a stabilization splint for the management of TMDs, combined with a structured counseling protocol delivered by the assigned dentist.

SUMMARY:
This prospective, longitudinal study investigates the influence of dentists' personality traits on patient-reported outcomes among individuals with temporomandibular disorders (TMDs) undergoing splint therapy. Dentists are assessed using the Big Five Inventory-2 Short Form (BFI-2-S), and patients are randomly assigned to them. Key outcomes measured six months after treatment include patient-centered communication, treatment satisfaction, adherence to splint therapy, and changes in psychological distress using validated scales such as the Patient-Centered Communication Scale (PCCS), a structured satisfaction questionnaire, and the DASS-10. The study explores whether traits such as conscientiousness, agreeableness, extraversion, openness, and emotional stability are associated with better patient outcomes in TMD care. This research aims to enhance patient-centered treatment by integrating personality-informed clinical practice and tailored communication strategies.

DETAILED DESCRIPTION:
Temporomandibular disorders are multifactorial conditions often accompanied by psychological distress, chronic pain, and functional limitations. While splint therapy remains a common conservative intervention, patient adherence and satisfaction with treatment can vary widely and are often influenced by interpersonal dynamics between provider and patient.

Emerging literature in medicine and dentistry suggests that provider personality traits play a critical role in shaping communication style, patient engagement, and ultimately clinical outcomes. However, few studies have systematically examined this relationship within dental practice, particularly in the management of TMDs.

This study adopts a prospective, randomized design. Thirty dentists treating TMD patients are assessed for their personality traits using the BFI-2-S, which evaluates five core dimensions: conscientiousness, agreeableness, extraversion, openness, and negative emotionality. Three hundred TMD patients are randomly assigned to one of the participating dentists and undergo a standardized treatment protocol involving splint therapy. Dentists follow a structured communication and counseling framework aimed at enhancing the quality of interaction and patient education.

Patient outcomes are assessed at baseline and after six months of therapy. The key outcomes include:

Quality of doctor-patient communication, measured using the PCCS,

Treatment satisfaction using a structured questionnaire,

Adherence to splint therapy (hours/day and days/week),

Psychological well-being measured by the DASS-10.

Statistical analyses include correlation to assess the association between dentist personality traits and patient outcomes.

This study has the potential to uncover meaningful links between provider personality and clinical success in TMD management. Results may guide the development of more effective communication protocols, inform training and self-awareness initiatives for dental professionals, and promote patient-centered care grounded in both technical and interpersonal excellence.

ELIGIBILITY:
Eligibility criteria for dentists included:

* Had at least two years of clinical experience in the management of TMDs.
* Were actively involved in the clinical care of TMD patients at the time of the study.
* Willingness to participate and complete the BFI-2-S personality assessment.

Eligibility criteria for patients included:

Inclusion Criteria:

* Diagnosed with TMDs according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) guidelines, specifically disc displacement with reduction.
* Exhibiting symptoms of stress or anxiety, as identified by the baseline DASS-10 screening.
* Prescribed occlusal splint therapy as part of their treatment regimen.

Exclusion Criteria:

* Cognitive impairments.
* Psychiatric conditions other than anxiety or depression.
* Any condition that could impair the patient's ability to provide informed consent or accurately complete self-report questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included adult patients diagnosed with TMDs seeking care at the oral and maxillofacial surgery department of Faculty of dentistry, Mansoura university. All patients were eligible for splint therapy and were randomly assigned to postgraduate dentists with advanced clinical training in TMD management. Dentists were with advanced training in TMD management. Participants were followed for six months after the initiation of treatment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Patient-Centered Communication Score (PCCS) | 6 months post-treatment
  Patient-centered communication was assessed using the validated Patient-PCCS. This self-reported measure evaluates the quality of dentist-patient communication from the patient's perspective, including aspects such as empathy, clarity, and involvement in decision-making. Scores range from low to high, with higher scores indicating more patient-centered communication. The outcome is used to determine the influence of dentist personality traits on perceived communication quality.

SECONDARY OUTCOMES:
Patient Satisfaction with Treatment | 6 months post-treatment
  Patient satisfaction was measured using a structured questionnaire developed to assess overall satisfaction with the treatment process, fulfillment of expectations, and perceived treatment effectiveness. Responses were scored on a Likert scale, with higher scores indicating greater satisfaction.
Adherence to Splint Therapy | 6 months post-treatment
  Patient adherence was assessed using two self-reported indicators: (1) average number of hours per day the splint was worn, and (2) number of days per week the splint was used consistently. Higher scores reflect better adherence.
Change in Psychological Distress (DASS-10 Score) | Baseline and 6 months post-treatment
  Psychological distress was measured using the 10-item Depression, Anxiety, and Stress Scale (DASS-10). The change in score from baseline to 6-month follow-up reflects improvement or worsening of psychological wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Soaad Tolba Badawy, Lecturer, Oral Surgery, MU, Principal Investigator — Faculty of dentistry, Mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided